CLINICAL TRIAL: NCT05010616
Title: The Influence of Showing Patients the Three-dimensional Digital Simulation of Their Teeth Alignment Produced by Orthodontic Treatment With Fixed Appliance on Their Expectations and Satisfaction
Brief Title: Evaluating the Influence of Showing Patients Their Predicted Teeth Alignment on Their Expectations and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-Ortho-07-2021
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Crowding, Tooth
Keywords: Crowding; Simulation; Prediction; Expectation; Satisfaction; Three-dimensional set up
MeSH Terms: conditions — Malocclusion; Crowding; Personal Satisfaction | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three-dimensional digital simulation with fixed appliance (Experimental): The records will be obtained at the first visit, which will be one week before placing brackets. At the second visit, the orthodontic appliances will be applied; then assessments will be taken after 15 minutes of showing the patient the digital simulation of their teeth alignment at the end of orthodontic treatment.
  Interventions: Device: Fixed orthodontic appliances

INTERVENTIONS:
Device: Fixed orthodontic appliances — Visual presentation of patient's predicted teeth alignment at the end of orthodontic treatment:
  Presenting predicted teeth alignment after orthodontic treatment to patients before treatment starts, by using photos and videos of dental digital set-up.
  Predicted teeth alignment can be described as: well-leveled and aligned patient's dental arches, well engaged posterior teeth and normal frontal teeth relationships.

SUMMARY:
Patients who have moderate crowding will be treated in this study. The efficacy of showing the predicted alignment of patient's teeth at the end of orthodontic treatment previously to treatment on their expectations from orthodontic treatment and their satisfaction with their teeth alignment will be assessed.

DETAILED DESCRIPTION:
It is known that most patients expect that orthodontic treatment will improve their appearance which increases their confidence and self-esteem level.

The ability to approach patient's expectations to reality is crucial to making them reasonable and to improve patient's satisfaction with treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Class I malocclusion with moderate crowding (between 4-6 mm of tooth-size-arch-length-discrepancy).
* Good oral hygiene and periodontal health.
* No severe skeletal discrepancy.
* Normal proclination for the upper and lower incisors.

Exclusion Criteria:

* Bimaxillary dentoalveolar severe protrusion.
* Need for extraction.
* Previous orthodontic treatment.
* Subject with psychological abnormalities.
* congenitally missing or extracted teeth (except for the third molars).
* history of previous trauma to the maxillofacial region or surgical interventions.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Change in patient's expectation towards teeth alignment: | T0: 1 week before placing brackets, T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment
  Patients will be asked: Do you expect the orthodontic treatment to straighten your teeth? Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not expected. Grades 1-3 = less expected. Grades 4-6 = average expected. Grades 7-9 = highly expected. Grade 10 = most expected.
Change in patient's expectation towards smile improvement | T0: 1 week before placing brackets, T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment
  Patients will be asked: Do you expect the orthodontic treatment to produce a better smile? Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not expected. Grades 1-3 = less expected. Grades 4-6 = average expected. Grades 7-9 = highly expected. Grade 10 = most expected.
Change in patient's expectation towards chewing improvement | T0: 1 week before placing brackets, T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment
  Patients will be asked: Do you expect the orthodontic treatment to make it easier to eat? Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not expected. Grades 1-3 = less expected. Grades 4-6 = average expected. Grades 7-9 = highly expected. Grade 10 = most expected.
Change in patient's expectations towards speech improvement | T0: 1 week before placing brackets, T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment
  Patients will be asked: Do you expect the orthodontic treatment to make it easier to speak? Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not expected. Grades 1-3 = less expected. Grades 4-6 = average expected. Grades 7-9 = highly expected. Grade 10 = most expected.
Change in patient's expectations towards oral hygiene improvement | T0: 1 week before placing brackets, T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment
  Patients will be asked: Do you expect the orthodontic treatment to make it easier to keep your teeth clean? Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not expected. Grades 1-3 = less expected. Grades 4-6 = average expected. Grades 7-9 = highly expected. Grade 10 = most expected
Change in patient's expectations towards getting a better career | T0: 1 week before placing brackets, T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment
  Patients will be asked: Do you expect the orthodontic treatment to improve your chance of a good career? Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not expected. Grades 1-3 = less expected. Grades 4-6 = average expected. Grades 7-9 = highly expected. Grade 10 = most expected.
Change in patient's expectations towards getting a better social confidence | T0: 1 week before placing brackets, T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment
  Patients will be asked: Do you expect the orthodontic treatment to give you confidence socially? Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not expected. Grades 1-3 = less expected. Grades 4-6 = average expected. Grades 7-9 = highly expected. Grade 10 = most expected.
  Scores of questions 1-2-3-4-5-6-7 will be summed to obtain total expectation's score.
  Questionnaires applied by patients at (T0) and (T1) will be compared by:
  * Comparing each question individually between T0 and T1.
  * Comparing questionnaire's overall score between T0 and T1.
Changes in patient's satisfaction with teeth appearance | T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment, T2: at the end of treatment after removing brackets
  Patients will be asked: Are you satisfied with your teeth appearance? Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not satisfied. Grades 1-3 = less satisfied. Grades 4-6 = average satisfaction. Grades 7-9 = highly satisfied. Grade 10 = most satisfied
Changes in patient's satisfaction with frontal teeth relationship | T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment, T2: at the end of treatment after removing brackets
  Patients will be asked: express your satisfaction with your frontal teeth relationship? Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not satisfied. Grades 1-3 = less satisfied. Grades 4-6 = average satisfaction. Grades 7-9 = highly satisfied. Grade 10 = most satisfied
Changes in patient's satisfaction level with teeth alignment | T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment, T2: at the end of treatment after removing brackets
  Patients will be asked: express your satisfaction with teeth alignment. Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not satisfied. Grades 1-3 = less satisfied. Grades 4-6 = average satisfaction. Grades 7-9 = highly satisfied. Grade 10 = most satisfied
Changes in patient's satisfaction level with teeth engagement | T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment, T2: at the end of treatment after removing brackets
  Patients will be asked: express your satisfaction with teeth engagement. Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not satisfied. Grades 1-3 = less satisfied. Grades 4-6 = average satisfaction. Grades 7-9 = highly satisfied. Grade 10 = most satisfied
Patient's overall satisfaction level with his teeth alignment following checking the predicated plan | T1: patient's second visit to clinician to begin the orthodontic treatment and after 15 minutes of showing patient the digital simulation of their teeth alignment at the end of orthodontic treatment
  Patients will be asked: express your overall satisfaction with your teeth after watching your predicted teeth alignment.
  Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10.
  Grade 0 = not satisfied. Grades 1-3 = less satisfied. Grades 4-6 = average satisfaction. Grades 7-9 = highly satisfied. Grade 10 = most satisfied.
Patient's overall satisfaction with his teeth at the end of orthodontic treatment | T2:at the end of orthodontic treatment after removing brackets] Patients will be asked: express your overall satisfaction with your teeth at the end of treatment.
  Question will be answered on paper using the Visual Analogue Scale (VAS) with grades from 0 to 10. Grade 0 = not satisfied. Grades 1-3 = less satisfied. Grades 4-6 = average satisfaction. Grades 7-9 = highly satisfied. Grade 10 = most satisfied
  Scores of questions 7-8-9-10-11-12 will be summed to obtain total expected satisfaction's score.
  Scores of questions 7-8-9-10-11-13 will be summed to obtain total eventual satisfaction's score.
  Questionnaires applied by patients at (T1) and (T2) will be compared by:
  * Comparing each question individually between T1 and T2.
  * Comparing questionnaire's overall score between T1 and T2.

CONTACTS AND LOCATIONS:
Overall Officials: Abd Alrahman Qusaibati, DDS, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental; Kinda sultan, DDS,MSc,PhD, Study Chair — Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grunheid T, Loh C, Larson BE. How accurate is Invisalign in nonextraction cases? Are predicted tooth positions achieved? Angle Orthod. 2017 Nov;87(6):809-815. doi: 10.2319/022717-147.1. Epub 2017 Jul 7. PMID 28686090
- [Background] Hadadpour S, Noruzian M, Abdi AH, Baghban AA, Nouri M. Can 3D imaging and digital software increase the ability to predict dental arch form after orthodontic treatment? Am J Orthod Dentofacial Orthop. 2019 Dec;156(6):870-877. doi: 10.1016/j.ajodo.2019.07.009. PMID 31784021
- [Background] Izhar A, Singh G, Goyal V, Singh R, Gupta N, Pahuja P. Comparative Assessment of Clinical and Predicted Treatment Outcomes of Clear Aligner Treatment: An in Vivo Study. Turk J Orthod. 2019 Dec 1;32(4):229-235. doi: 10.5152/TurkJOrthod.2019.19019. eCollection 2019 Dec. PMID 32110468
- [Background] Noroozi H, Djavid GE, Moeinzad H, Teimouri AP. Prediction of arch perimeter changes due to orthodontic treatment. Am J Orthod Dentofacial Orthop. 2002 Dec;122(6):601-7. doi: 10.1067/mod.2002.128213. PMID 12490870
- [Background] Buschang PH, Ross M, Shaw SG, Crosby D, Campbell PM. Predicted and actual end-of-treatment occlusion produced with aligner therapy. Angle Orthod. 2015 Sep;85(5):723-7. doi: 10.2319/043014-311.1. Epub 2014 Nov 5. PMID 25372019
- [Derived] Kusaibati AM, Sultan K, Hajeer MY, Burhan AS, Alam MK. Adult patient expectations and satisfaction: Can they be influenced by viewing the three-dimensional predicted outcome before fixed orthodontic treatment of dental crowding? J World Fed Orthod. 2023 Dec;12(6):269-279. doi: 10.1016/j.ejwf.2023.08.005. Epub 2023 Sep 28. PMID 37777351